CLINICAL TRIAL: NCT03590158
Title: The Metabolic Impacts of Time-restricted Feeding in Men at High Risk of Type 2 Diabetes
Brief Title: Time RestrIcted Feeding For Improving Diabetes Risk (TRIFFID)
Acronym: TRIFFID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Adelaide (Other)
Collaborators: University of South Australia (Other); Salk Institute for Biological Studies (Other)
Responsible Party: Principal Investigator, A/Prof Leonie Heilbronn, A/Prof, University of Adelaide
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R20180320
Record Dates: First submitted 2018-07-12; First posted 2018-07-18 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Type2 Diabetes; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRF (Experimental): Participants will follow their regular diet for two weeks before 3-day lead-in food prior to the metabolic testing at visit 0. Participants will then be instructed to eat their habitual diet only within a 10-hour time frame each day for 8 weeks. Participants may self-select the precise window that best suits their lifestyles, however any food and drink must be consumed by 7:30pm.
  Interventions: Behavioral: TRF

INTERVENTIONS:
Behavioral: TRF — Participants will be instructed to consume their habitual diet within a self-selected 10 hour period every day.

SUMMARY:
This study will explore the effects of eight weeks of time-restricted feeding (TRF) on body weight and composition, glycaemic control, 24-hour glucose profiles, glucoregulatory hormones, and cardiovascular risk in men at high risk of type 2 diabetes. The investigators hypothesise that 8 weeks of TRF will reduce body weight, improve body composition, improve glycaemic control and blood lipid profiles. The potential mechanism will be explored in terms of the changes in gene expression patterns and multi-omics level (e.g., adipose tissue transcriptome, blood proteome).

DETAILED DESCRIPTION:
Following a 2 week baseline monitoring phase (food intake by smartphone APP, activity by accelerometer, glucose by continuous glucose monitor), participants will attend the metabolic clinic for testing (visit 0). Body weight, body composition (by DEXA), and blood pressure will be assessed. Blood and adipose tissue samples will be collected over 24-hour period for assessment of glucose, insulin, glucoregulatory hormones, blood lipids and adipose tissue transcriptome. Glucose and insulin responses to a standardised breakfast will be measured. All food will be provided for 3 days prior to the metabolic visit. Following visit 0, participants will be instructed to eat only within a 10-hour time frame each day for 8 weeks. Participants may self-select the precise window that best suits their lifestyles, however any food and drink must be consumed at least 3 hours prior to their usual bedtime. 24-hour glucose profiles, activity and food intake will be measured again at week 6-8. At the end of the 8 weeks, participants will return for a follow-up metabolic visit, identical to that at visit 0, except foods are provided with the 10h time frame.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference ≥94 cm
* Weight-stable (< 5 % fluctuation in their body weight for past 6-months at study entry)

Exclusion Criteria:

* Personal history and/or diagnosis of: diabetes, cancer, major psychiatric disorders, liver disease, gastro-intestinal surgery or disease (including malabsorption), eating disorders, anaemia, insomnia, cardiovascular disease deemed unstable by the study physician.
* use of prescribed or non-prescribed medications which may affect energy metabolism, gastrointestinal function, body weight or appetite, sleep (e.g: domperidone and cisapride, anticholinergic drugs (e.g.: atropine), metoclopramide, orlistat, thyroid medications, diuretics, glucocorticoids, sex steroids, metformin, dipeptidyl peptidase-IV inhibitors, melatonin)
* recent weight change in past 3 months (> 5% current body weight)
* individuals who regularly perform high intensity exercise (>2 week)
* current intake of > 140g alcohol/week
* current smokers of cigarettes/cigars/marijuana/e-cigarettes/vaporisers
* current intake of any illicit substance
* unable to comprehend study protocol
* currently performing shift work
* has undertaken, or is planning to undertake, trans meridian travel during the study period, or the preceding 60 days
* do not own a smartphone
* eats for less than a 12-hour period per day

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2019-06-29 (Actual)

PRIMARY OUTCOMES:
Glycaemia | 2.5 hours
  Change in postprandial glucose (iAUC) following a standard breakfast

SECONDARY OUTCOMES:
Insulin | 2.5 hours
  Change in fasting and postprandial insulin following a standard breakfast.
HbA1c | 8 weeks
  Change in HbA1c
Body weight | 8 weeks
  Change in body weight
Body composition | 8 weeks
  Change in body fat mass and fat free mass
Waist and hip circumference | 8 weeks
  Change in waist and hip circumference
24-hour glucose profile | 8 weeks
  Change in 24-hour glucose profiles assessed by continuous glucose monitoring
Blood pressure | 8 weeks
  Changes in systolic blood pressure and diastolic blood pressure
Blood lipids | 8 weeks
  changes in blood lipid profile (total cholesterol, HDL-, LDL- cholesterol and triglycerides)
Non-esterified fatty acid (NEFA) | 8 weeks
  Change in non-essential fatty acid (NEFA)
Plasma gastrointestinal (GI) hormones | 8 weeks
  Changes in concentration of fasting and postprandial GI hormones in plasma (ghrelin, glucagon-like peptide-1, glucose-dependent insulinotropic polypeptide, peptide YY) following a standard breakfast.
Plasma cortisol | 8 weeks
  Changes in concentration of cortisol in hourly plasma samples assessed from 6am to 12pm.
Plasma Melatonin | 8 weeks
  Changes in dim light melatonin onset (DLMO) assessed from 5pm to 3am
Adipose tissue transcriptome | 8 weeks
  A subset will be measured for the change in the adipose tissue transcriptome in 6-hourly samples by RNA-sequencing. The data analysis including but not limited to the changes in numbers of genes oscillated in a diurnal manner, and pathway analysis.
Evening glycaemia | 8 weeks
  An ancillary study will be performed to measure the changes in the concentration of plasma glucose, insulin and GI hormones (ghrelin, glucagon-like peptide-1, glucose-dependent insulinotropic polypeptide, peptide YY) following a standard evening meal.
Physical activity and sleep | 8 weeks
  An ancillary study will measure the changes in sleep and physical activity monitored by a wrist actigraph for 14 days.
Food intake and meal timing | 8 weeks
  An ancillary study will measure the changes in food intake and meal timing as recorded via a photography based smartphone App over 2 weeks. The analysis of the App data including but not limited to eating duration at baseline, changes in eating duration after intervention, calorie distribution throughout the day, meal frequency, meal intervals, and macronutrients intake.
Continuous glucose monitoring | 8 weeks
  An ancillary study will measure the changes in glucose level by CGM for 14 days. Daily glucose patterns including free habitual diet, 3-day lead-in food will be measured separately. The analysis of the CGM data including but not limited to assess the mean amplitude of glycaemic excursions (MAGE), continuous overall net glycaemic action (CONGA), mean glucose concentrations.
Objective sleep | 8 weeks
  Changes in objective sleep status measured by laboratory polysomnography (PSG).

OTHER OUTCOMES:
Hair follicle clock gene expression | 8 weeks
  Changes in the circadian pattern of clock gene expression in hair follicles.
Resting metabolic rate | 8 weeks
  A subset of participants will be examined for the changes in resting metabolic rate and respiratory quotient.
Metagenomics and metabolomics | 8 weeks
  Changes in metagenome and metabolome in a subset of participants will be assessed in faeces by shotgun metagenomics sequencing and metabolites analysis. The data analysis including but not limited to the function and composition of the gut microbiota, and faecal bile acids.
Plasma proteome | 8 weeks
  Plasma proteome will be assessed by mass-spectrometry driven analysis. The data analysis including but not limited to the changes in numbers of proteins oscillated in a diurnal manner, and pathway analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Leonie Heilbronn, PhD, Principal Investigator — University of Adelaide
Locations (1):
- University of Adelaide, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No